CLINICAL TRIAL: NCT06262204
Title: Clinical and Radiological Comparison of Hallux Valgus Correction Using the Metal Screw or the Human Allogeneic Cortical Bone Screw, a Prospective Study
Brief Title: Hallux Valgus Correction Using the Metal Screw or the Human Allogeneic Cortical Bone Screw (Shark Screw).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Forian Wenzel-Schwarz, principal investigator, Orthopedic Hospital Vienna Speising
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hallux Shark Screw(R)
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hallux Valgus
Keywords: Hallux Valgus; human allogeneic cortical bone screw; Shark Screw®; HVA; IMA; AOFAS; time to union; union rate; FFI
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant
Masking Description: does get the information only after 2 years at the end of teh study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Other): standard surgery with metal screw
  Interventions: Procedure: Hallux Valgus Treatment with metal screw
- Shark Screw® group (Experimental): new surgical procedure with human allogeneic cortical bone screw
  Interventions: Procedure: Hallux Valgus Treatment with Shark Screw®

INTERVENTIONS:
Procedure: Hallux Valgus Treatment with Shark Screw® — This is a prospective, randomised study in which hallux valgus is corrected by means of a chevron/kin surgery technique using metal screws or human allogenic cortical bone screws (Shark Screw®, Surgebright, Lichtenberg, Austria). X-rays are taken before the operation at 6 weeks, three, six and twelve months after the operation. The X-ray images provide information on whether bony degeneration has taken place. In addition, the American Orthopaedic Foot & Ankle Society (AOFAS) hallux score, FFI score, hallux valgus angle (HVA) and intermetatarsal angle (IMA) are determined. These data are collected preoperatively and 4 weeks (HVA and IMA), six and twelve months postoperatively in order to rule out a change in the HVA and IMA and to document the changes in the AOFAS/FFI.
  Arms: Shark Screw® group
Procedure: Hallux Valgus Treatment with metal screw — This is a prospective, randomised study in which hallux valgus is corrected by means of a chevron/kin surgery technique using metal screws or human allogenic cortical bone screws (Shark Screw®, Surgebright, Lichtenberg, Austria). X-rays are taken before the operation at 6 weeks, three, six and twelve months after the operation. The X-ray images provide information on whether bony degeneration has taken place. In addition, the American Orthopaedic Foot & Ankle Society (AOFAS) hallux score, FFI score, hallux valgus angle (HVA) and intermetatarsal angle (IMA) are determined. These data are collected preoperatively and 4 weeks (HVA and IMA), six and twelve months postoperatively in order to rule out a change in the HVA and IMA and to document the changes in the AOFAS/FFI.
  Arms: conventional group

SUMMARY:
The goal of this clinical trial is to compare the treatment of Hallux Valgus using the conventional method (metal screw) with the new method (human allogeneic cortical bone screw (Shark Screw®) in adult patients with confirmed Hallux Valgus.

The main questions it aims to answer are:

Can the new method obtain comparable results as the conventional method in regard to union rate and time to union? Are the number of complications lower with the new method? Participants will be operated either with the metal screw or with the Shark Screw®. The assignment to the groups is randomized.

DETAILED DESCRIPTION:
The planned prospective study will investigate whether the use of the human allogenic cortical bone screw (Shark Screw® leads to comparable results in the union rate and the prevention of recurrences as with metal screws. Furthermore, it will be investigated whether rotational stability is possible with the bone screw. The measurement of the HVA angle and the IMA angle should provide information on whether the correction is stable over time. A comparison of the AOFAS forefoot score before and after the operation for both methods is a further measure to check whether the human allogenic cortical bone screw can deliver similar results.

Initial studies on the use of the allogenic bone screw in hand and foot surgery show particularly good integration behavior of the human allogenic cortical bone screw . A retrospective study by Hanslik-Schnabel et al has shown initial positive results in the treatment of hallux rigidus. In addition, a gait analysis is performed pre- and postoperatively to provide information on possible differences between the two groups in the context of 3D gait analysis/pedobarography and is also matched with another healthy cohort.

At the preoperative time point and after 12 and 24 months, a 3D gait analysis with a foot model is conducted to record the joint kinematics and kinetics. In the study by Canseco et al. , the proximal gait pattern changes remained unchanged. Hwang reported hyper-external rotation in the subtalar joint, excessive eversion in the subtalar joint, and lack of movement in the hallux MP joint in the terminal standing phase.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 85
* confirmed Hallux Valgus

Exclusion Criteria:

* <18 years and >85 years
* Known underlying oncological disease
* Pregnant women or breastfeeding mothers
* Alcohol and drug abuse
* Foreseeable compliance problems
* Foreseeable loss of responsibility as a study doctor
* Neoplastic diseases
* Active osteomyelitis
* Ulcerations in the area of the skin of the surgical site
* Immunosuppressive medication that cannot be discontinued

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical result of Hallux Valgus treatment | 2 years
  The primary objective of the study is the longitudinal evaluation of clinical outcomes (pain, appearance) over 2 years after hallux correction using a human, allogenic, bone screw or metal screw.

SECONDARY OUTCOMES:
radiological (bony union)result of Hallux Valgus treatment | 1 years
  The secondary aim of the study is the longitudinal evaluation of the radiological results over one year after hallux correction using a human, allogenic, bone screw or metal screw compared to pre-surgery values.
change in forefoot-American Orthopaedic Foot and Ankle Society (AOFAS) | 2 years
  The change in forefoot-AOFAS will be evaluated, between groups and in comparison to pre-surgery
Hallux-Valgus angle (HVA) change | 2 years
  Comparison of HVA pre-surgery and after 6, 12 and 24 months after surgery, between groups and in comparison to pre-surgery data
gait analysis | 2 years
  Number of patients with normal gait in the two groups and in comparison to a healthy cohort
Intermetatarsal angle (IMA) change | 2 years
  Comparison of IMA pre-surgery and after 6, 12 and 24 months after surgery, between groups and in comparison to pre-surgery data

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wenzel-Schwarz, MD, Principal Investigator — Orthopädisches Spital Speising
Locations (1):
- Abteilung für Kinderorthopädie und Fußchirurgie Orthopädisches Spital Speising, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Due to sensitivity of Data